CLINICAL TRIAL: NCT04787055
Title: A Study to Examine the Performance of a Hearing Aid Transducer During Typical, In-field Use
Brief Title: In Field Performance of a Hearing Aid Transducer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sonova AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SRF-61
Record Dates: First submitted 2021-01-28; First posted 2021-03-08 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2022-05

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Receiver in the canal hearing instrument 3 month (Experimental): Group of subjects who will get the receiver in the canal hearing instrument and wear for period of three months.
  Interventions: Device: Receiver-in-canal hearing instrument
- Receiver in the canal hearing instrument 6 month (Experimental): Group of subjects who will get the receiver in the canal hearing instrument and wear for period of six months.
  Interventions: Device: Receiver-in-canal hearing instrument

INTERVENTIONS:
Device: Receiver-in-canal hearing instrument — Receiver-in-canal hearing instrument

SUMMARY:
Study participants will be fit with previously released receiver-in-canal (RIC) hearing instruments. Participants will be asked to wear the instruments in their daily life for a minimum of 3 months, but have the option to continue to wear devices for six months.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate sensorineural hearing loss
* Adult

Exclusion Criteria:

* Inability or unwillingness to wear study devices for extended period of time.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Phonak Audiology Research Center, Aurora, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Receiver in the Canal Hearing Instrument 3 Month: Group of subjects who will get the receiver in the canal hearing instrument and wear for three months.
- Receiver in the Canal Hearing Instrument 6 Month: Group of participants who will get the receiver in the canal hearing instrument and wear for six months.
Period: Overall Study
Arm/Group | Receiver in the Canal Hearing Instrument 3 Month | Receiver in the Canal Hearing Instrument 6 Month
Started | 18 | 17
Completed | 15 | 11
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Receiver in the Canal Hearing Instrument 3 Month: Group of subjects who will get the receiver in the canal hearing instrument for a 3 month period.
- Receiver in the Canal Hearing Instrument 6 Month: Group of subjects who will get the receiver in the canal hearing instrument for a 6 month period.
- Total: Total of all reporting groups
Arm/Group | Receiver in the Canal Hearing Instrument 3 Month | Receiver in the Canal Hearing Instrument 6 Month | Total
Number analyzed (Participants) | 18 | 17 | 35
Age, Continuous [Mean (Full Range); unit: years] | 73 [55 to 87] | 72 [55 to 87] | 72.5 [55 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 11 | 11 | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Subjective Satisfaction of Hearing Aid Performance in Noisy Environments
Description: Subject rates how satisfied they are with performance of hearing aid while listening in noisy environments. Ratings range from 1 (very dissatisfied) to 5 (very satisfied) with 3 = Neither satisfied or dissatisfied.
Time Frame: Three months after initial appointment
Population: Participants who answered the question "How satisfied are you with the performance of the hearing aids in noisy environments?" after 3 months of wearing devices.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Receiver in the Canal Hearing Instrument 3 Month
Number analyzed (Participants) | 15
score on a scale | 3.86 [2 to 5]

2. Primary Outcome: Subjective Satisfaction of Hearing Aid Performance in Noisy Environments
Description: as for outcome 1
Time Frame: Six months after initial appointment
Population: Participants who wore device for six months and answered the question "How satisfied are you with the performance of the hearing aids in noisy environments?" at the end of the six months.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Receiver in the Canal Hearing Instrument 6 Month
Number analyzed (Participants) | 11
score on a scale | 2.73 [2 to 5]

3. Primary Outcome: Subjective Satisfaction of Hearing Aid Performance While Listening to Streamed Media
Description: Subject rates how satisfied they are with performance of hearing aid when listening to a streamed signal (i.e. music, video, etc.) Ratings range from 1 (very dissatisfied) to 5 (very satisfied) with 3 = Neither satisfied or dissatisfied.
Time Frame: Three months after initial appointment
Population: Participants who wore devices for three months and who answered the question at the end of the 3 months "How satisfied were you with the performance of the hearing aid when streaming?"
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Receiver in the Canal Hearing Instrument 3 Month
Number analyzed (Participants) | 15
score on a scale | 4.67 [2 to 5]

4. Primary Outcome: Subjective Satisfaction of Hearing Aid Performance While Listening to Streamed Media
Description: as for outcome 3
Time Frame: Six months after initial appointment
Population: Participants who wore devices for 6 months and who answered the question at the end of the 6 months "How satisfied were you with the performance of the hearing aid when streaming?"
Measure: Mean (Full Range); unit: score on a scale
Groups:
- Receiver in the Canal Hearing Instrument 6 Months: Group of subjects who will get the receiver in the canal hearing instrument for a 6 month period.
Arm/Group | Receiver in the Canal Hearing Instrument 6 Months
Number analyzed (Participants) | 11
score on a scale | 4.36 [4 to 5]

ADVERSE EVENTS:
Time Frame: Three months for participants who were in the group assigned devices for three months, and six months for the participants who were in group assigned devices for six months.
Arm/Group | Receiver in the Canal Hearing Instrument 3 Month | Receiver in the Canal Hearing Instrument 6 Month
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/17
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/17
Other Adverse Events (participants affected / at risk) | 0/18 | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Receiver in the Canal Hearing Instrument 3 Month (N=18) | Receiver in the Canal Hearing Instrument 6 Month (N=17)
Unanticipated death (Renal and urinary disorders) | 0 (0) | 1 (1) — Participant was diagnosed with bladder cancer during the course of the study and passed away from bladder cancer. This was unrelated to study procedure or study devices.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-02-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT04787055/Prot_001.pdf